CLINICAL TRIAL: NCT03578094
Title: Impact of Feeding Patterns on Adiposity and Cardiometabolic Markers in Baby and Mother: A Prospective Cohort Study
Brief Title: Mother and Infant Study Cohort (MISC)-
Status: Completed | Type: Observational
Sponsor: University of Sharjah (Other)
Collaborators: Al Jalila Foundation (Unknown)
Responsible Party: Principal Investigator, Hadia Radwan, Assistant Professor, University of Sharjah
Other Study IDs: 1501057003-P
Record Dates: First submitted 2018-05-02; First posted 2018-07-05 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-06

CONDITIONS: Adiposity, Breast Feeding
Keywords: cohort; Noncommunicable diseases; pregnancy; infant; cognition; United Arab Emirates; gestational diabetes
MeSH Terms: conditions — Obesity; Breast Feeding; Noncommunicable Diseases; Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breastmilk samples, blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to explore breastfeeding and complementary feeding practices of mothers in the United Arab Emirates (UAE) and its relation to the early life determinants of obesity and non-communicable diseases (NCDs). This research study will follow a prospective cohort approach. Two hundred and fifty mother-infant pairs will be followed for 18 months.

The hypothesis of this research study is that exclusive breastfeeding of the infant will provide potential protective effect against cardiometabolic risk factors. This study will also hypothesize that mothers who exclusively breastfeed their newborns would experience greater postpartum weight and body fat loss than mothers who are not breastfeeding.

DETAILED DESCRIPTION:
United Arab Emirates(UAE) is facing two critical situations: high incidence of obesity and chronic diseases and suboptimal infant feeding practices as reported by the Ministry of Health in the UAE. So early identification of preventive markers of cardiometabolic risk factors in breast milk is important for developing early intervention strategies to optimize health care for individuals and communities especially in countries suffering from high rates of obesity and chronic diseases such as the UAE.

The purpose of this study is to prospectively follow up with the mothers and their infants (from 0-18months of infants age). It will explore breastfeeding and complementary feeding practices of mothers in UAE and its relation to the early life determinants of obesity and non-communicable diseases (NCDs). It will examine the components of human milk which might offer a protective benefit against obesity and its health consequences in infancy. It will also evaluate the feeding practices of the mothers and her nutritional status and relates it to their infants' growth and development.

It is expected that this research study will fill an important knowledge gap in the understanding of the feeding practices of mothers and its relation to early-life determinants of obesity and other chronic diseases in the UAE.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women:

  * Emirate nationality or Arab expatriate
  * Age: 19-40 years
  * Singleton pregnancy
  * Within the third trimester of pregnancy (27-42 weeks of gestation)
  * Free of chronic diseases (diabetes, hypertension, kidney disease, cancer, or other chronic diseases), autoimmune disorders, or infections with the human immunodeficiency virus, or hepatitis in preconception

Exclusion Criteria:

* Multiple pregnancies (pregnant with two or more fetuses)
* High-risk pregnancy or pre-eclampsia
* History of chronic diseases
* Preterm (<37 weeks of gestation) or late-term (>42 weeks of gestation) infants
* Congenital diseases or any health condition that could deter breastfeeding

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The sample population is Emirati and Arab expatriate mothers, aged 19 to 40 years old; visiting Mother and Child Centers (MCH) and Primary Healthcare Centers (PHC) in Dubai and Sharjah.
  The selected mothers (who will be recruited during their 3rd trimester) were invited to participate in the study after being consented for their procedures and they will sign on the behalf of their babies
Sampling Method: Non-Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
relationship between exclusive breastfeeding and maternal serum levels of adiponectin | 18 months
  measuring the adiponectin level in the maternal serum at 6 months postpartum
relationships between maternal milk levels of adiponectin with infants serum levels of adiponectin | 18 months
  measuring the adiponectin level and in the infants serum and in the breast milk
Comparison of the infant adiponectin serum level in exclusive breastfeeding mothers versus mothers who do not exclusively breastfeed their infants | 18 months
  measuring the adiponectin serum level in the infants of exclusive breastfeeding group and other breastfeeding patterns
Association between duration of breastfeeding and mothers' anthropometric measurements(weight in kilograms and Height in meters ) | 18 months
  Measuring the weight in kilograms and height in meters weight and height will be combined to report BMI in kg/m^2 of the mothers at different timelines in relation to breastfeeding duration
Assessment of the anthropometric measurements (weight in kilograms and height in meters) of the mothers according to the breastfeeding patterns | 18 months
  Measuring the weight in kilograms and height in meters weight and height will be combined to report BMI in kg/m^2 of mothers at different timelines in relation to different breastfeeding patterns
relationship between exclusive breastfeeding and breast milk levels of adiponectin | 18 months
  measuring the adiponectin level in the breast milk at 6 months postpartum
Assessment of the anthropometric measurements of the infant according to the breastfeeding patterns | 18 months
  measuring the weight, height, mid upper arm circumference of the infant at different timelines in relation to the breastfeeding patterns

CONTACTS AND LOCATIONS:
Overall Officials: Hadia Radwan, PhD, Principal Investigator — University of Sharjah
Locations (1):
- Hadia Radwan, Sharjah city, Shajah, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after November 2018
Access Criteria: permission from the PI